CLINICAL TRIAL: NCT02125981
Title: A Prospective Randomized Double-blinded Clinical Trial About the Efficacy of Oral Limaprost Administration Following Surgery for Cervical Myelopathy
Brief Title: The Study About the Efficacy of Oral Limaprost After Surgery for Cervical Myelopathy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIMA_001
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Cervical Myelopathy
Keywords: limaprost alfadex; cervical myelopathy; surgery
MeSH Terms: interventions — limaprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Limaprost (Experimental): taking Limaprost α-Cyclodextrin Clathrate 1 Tablets (166.67 μg), three times per day
  Interventions: Drug: Limaprost
- Control (Placebo Comparator): taking placebo drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Limaprost — taking Limaprost α-Cyclodextrin Clathrate 1 Tablets (166.67 μg), three times per day
  Arms: Limaprost
Drug: Placebo — taking placebo drug
  Arms: Control

SUMMARY:
The limaprost alfadex can improve the surgical outcomes in patients with cervical myelopathy.

ELIGIBILITY:
Inclusion Criteria:

* Older than 20 years old
* Compressive cervical myelopathy, confirmed by MRI, including C1-C2 instability, ossification of posterior longitudinal ligament
* Plan to undergo cervical surgery for myelopathy
* JOA score less than 15 points
* Signed informed consent of patient or legal guardian

Exclusion Criteria:

* Infection or malignancy
* Taking Limaprost before surgery
* Pregnancy or expected to be pregnant or breast feeding
* severe cardiovascular, pulmonary, renal disease or distress, brain pathology
* any related coagulopathy
* any drug to cause bleeding tendency
* severe pain from other disease
* any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study
* patient cannot follow study protocol, for any reason

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Japanese Orthopedic Association (JOA) recovery rates | up to 12 months after operation
  JOA recovery rate = [(postoperative JOA score) - (preoperative JOA score)] / [(17-(preoperative JOA score)] x 100 (%).

SECONDARY OUTCOMES:
Visual Analog Pain Scale for neck pain | up to 12 months after operation
Neck disability index score | up to 12 months after operation
Japanese orthopaedic association Cervical Myelopathy Evaluation Questionnaire score | up to 12 months after operation
Questionnaire Short Form 12 | up to 12 months after operation
Japanese orthopaedic association score | up to 12 months after surgery
assessment of the efficacy of positron emission tomography (PET) | up to 12 months after operation
  The assessment of the efficacy of PET for prediction of drug (Limaprost) effect

CONTACTS AND LOCATIONS:
Overall Officials: Jin S. Yeom, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea